CLINICAL TRIAL: NCT04612270
Title: Quantification of Clinically Relevant Drug Induced Changes in HbO2 Affinity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1265/2020
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants for blood collection (Experimental): The blood samples of all participants will be treated equally according to the study protocol. No intervention in-vivo.
  Interventions: Other: Venous blood collection

INTERVENTIONS:
Other: Venous blood collection — Two venous blood collections in within one week. No drug-related intervention in-vivo.

SUMMARY:
The presented study is an experimental in-vitro study without intervention in-vivo. The effects of nitric oxide and prostacyclins, 5-hydroxymethylfurfural and alpha-ketoglutarate, volatile anaesthetics on haemoglobin oxygen (HbO2) affinity will be investigated in-vitro. Venous blood samples of 20 healthy young volunteers (10 female, 10 male) will be collected twice in the period of one week. Informed consent will be given. Every blood collection will be accompanied by a venous blood gas analysis. The blood samples will be transferred to the laboratory for in-vitro recording of the complete oxygen dissociation curve (ODC). A newly developed in-vitro method will be used. On the first study day the blood samples will be exposed to three different concentrations of nitric oxide during the measurement, followed by two different vapourized prostacyclins. In addition, different concentrations of 5-hydroxymethylfurfural and alpha-ketoglutarate will be given to the blood samples for ODC recording. On the second study day the dose dependent effects of three different volatile anaesthetics will be investigated by exposing the blood samples to these drug while the measurements. Following these ODC recordings, aliquots of the blood samples will be frozen and investigated for storage related changes in HbO2 affinity.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* ASA 1 (American Society of Anesthesiologists classification)

Exclusion Criteria:

* Any drug intake within 10 days prior to blood collection
* Smoking
* Haemoglobinopathy
* Acute inflammatory disease within 14 days prior to blood collection
* Pregnancy or breastfeeding
* Severe trauma or blood loss within 14 days prior to blood collection
* Participation in any other clinical study
* High altitude sojourn for several days (> 3,000 m) within four weeks prior to blood collection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 10 female and 10 male participants.
Enrollment: 22 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
P50 | One day
  Partial pressure of oxygen, at which 50% of haemoglobin is saturated with oxygen.

SECONDARY OUTCOMES:
Hill coefficient | One day
  Parameter describing the cooperativity of oxygen ligand binding to haemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ströhle, MD, Principal Investigator — MUI, Department of Anaesthesiology and Critical Care Medicine
Locations (1):
- Department of Anaesthesiology and Critical Care Medicine, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ronzani M, Woyke S, Mair N, Gatterer H, Oberacher H, Plunser D, Haller T, Strohle M, Rugg C. The effect of desflurane, isoflurane and sevoflurane on the hemoglobin oxygen dissociation curve in human blood samples. Sci Rep. 2022 Aug 10;12(1):13633. doi: 10.1038/s41598-022-17789-6. PMID 35948604